CLINICAL TRIAL: NCT00845689
Title: Study on the Potential Role of Intraoperative Hepatoprotection During Liver Resections
Brief Title: Prevention of Liver Damage During Liver Surgery
Acronym: LTR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Prof. Dr. Manfred Thiel, Department of Anaesthesiology of the Ludwig-Maximilians-University
Other Study IDs: LMU-202-LTR
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Liver Tumors
Keywords: liver surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Adenosine; Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): liver resection with Pringle + placebo
  Interventions: Drug: placebo; Procedure: Liver resection
- 2 (Active Comparator): liver resection with Pringle + adenosine preconditiong
  Interventions: Drug: adenosine; Procedure: Liver resection
- 3 (Active Comparator): liver resection with Pringle + adenosine pre- and postconditioning
  Interventions: Drug: adenosine; Procedure: Liver resection

INTERVENTIONS:
Drug: placebo — NaCl 0,9 %
  Arms: 1
Drug: adenosine — intravenous infusion of adenosine 0, 2 %
  Arms: 2
Drug: adenosine — intravenous infusion of adenosine 0,2 %
  Arms: 3
Procedure: Liver resection — Liver resection with Pringle maneuver

SUMMARY:
Liver damage as a consequnce of ischemia (I) and reperfusion (R) is known to harm the liver and could hence be a critical factor of the postoperative outcome of patients undergoing liver surgery. In order to protect the liver from ischemic damage following interventions such as the Pringle Maneuver, preconditioning has been successfully applied in various animal models as well as in humans. Since ischemia inevitably leads to cell hypoxia and subsequnet release of endogenuous metabolites, the investigators hypothesize that instead of brief periods of ischemia, the exogenuous infusion of purine analogues may also protect against subsequent prolonged periods of ischemia. Moreover, after reperfusion, the antiinflamamtory action of purine ananlogue infusion can further attenuated liver damage.

ELIGIBILITY:
Inclusion Criteria:

* elective resection of liver tumors
* age 18 to 80 years
* informed consent

Exclusion Criteria:

* chronic obstructive pulmonary disease
* heart insufficiency NYHA III-IV
* atrio-ventricular conductance blockage II. (Mobitz) or III. degree
* atrial fibrillation
* coronary heart disease (CCS III. or IV. degree)
* arterial hypertension
* acute renal failure
* increased intracranial pressure
* gout
* pregnancy

Age Groups: Child, Adult, Older Adult